CLINICAL TRIAL: NCT03438253
Title: Unwanted Penile Engorgement in Pediatric Patients Under Anesthesia: A Prospective Cohort Study to Discuss the Role of Anesthetic Technique and Other Common Contributing Factors.
Brief Title: Unwanted Penile Engorgement in Pediatric Patients Under Anesthesia.
Status: Completed | Type: Observational
Sponsor: Aligarh Muslim University (Other)
Responsible Party: Principal Investigator, MUAZZAM HASAN, Assistant Professor, Aligarh Muslim University
Other Study IDs: UWIPE
Record Dates: First submitted 2018-02-10; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Anesthesia; Functional
Keywords: Intraoperative penile engorgement; Anaesthesia; Urogenital surgery
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: spinal anaesthesia
  Other Names: sedation

SUMMARY:
Penile engorgement during intraoperative period is of rare occurrence however when do happens, leads to difficulty in performing and even cancellation of elective urogenital surgery. The mechanism behind intraoperative penile engorgement is complex and involves various factors. One common myth is that penile engorgement occurs only during spinal anaesthesia and not in general anaesthesia. In this study we intend to report the incidence and management of intraoperative penile engorgement in pediatric patients undergoing urogenital operations under spinal anesthesia with/without sedation over a period of one year. The pathophysiology and role of common contributing factors leading to intraoperative penile engorgement are also discussed.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist grade1 & 2
* Elective urogenital surgery of expected duration less than one hour

Exclusion Criteria:

* patients with local infection, coagulation abnormalities, expected duration of surgery >1 hour and spinal anomalies.
* parents of patient not giving consent for spinal anaesthesia.

Ages: 2 Years to 12 Years | Sex: Male
Age Groups: Child
Study Population: All ASA grade 1 & 2 pediatric patients having age between 2 to 12 years.
Enrollment: 386 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Intraoperative penile engorgement | sixty minutes from start of anaesthesia
  Incidence of intraoperative penile engorgement under anaesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Muazzam Hasan, MD, Principal Investigator — Assistant Professor